CLINICAL TRIAL: NCT05277155
Title: A Randomized, Controlled and Double-blinded Clinical Trial to Investigate the Efficacy and Safety of BEJO Red Ginger as an Adjuvant Therapy in COVID-19 Hospitalized Patients With Mild Symptoms
Brief Title: Trial to Study the Efficacy and Safety of BEJO Red Ginger in COVID-19 Patients With Mild Symptoms
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Research Center for Chemistry, National Research and Innovation Agency of Indonesia (Other Government)
Collaborators: National Research and Innovation Agency of Indonesia (Unknown); RSDC Wisma Atlet (Unknown); PT. Bintang Toedjoe (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 20-12-1505
Record Dates: First submitted 2022-03-04; First posted 2022-03-14 (Actual); Last update posted 2022-03-14 (Actual); Status verified 2022-03

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Intervention Model Description: patient will be randomized 1:1 to placebo with SOC and BEJO Red Ginger with standard of care (SOC).
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (BEJO Red Ginger Extract) (Experimental): 84 patients, dosage: BEJO Red Ginger Extract orally administrated 3 times a day each 15 mL plus the standard COVID-19 treatment as per hospital guideline with 2 hours interval time. (Time frame: from randomization to day 14 or until hospital discharge)
  Interventions: Dietary Supplement: BEJO Red Ginger Extract
- Control Group (Placebo) (Placebo Comparator): 84 patients, dosage: Placebo orally administrated 3 times a day each 15 mL plus the standard COVID-19 treatment as per hospital guideline with 2 hours interval time. (Time frame: from randomization to day 14 or until hospital discharge)
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: BEJO Red Ginger Extract — BEJO Red Ginger Extract ingredients:
  * Zingiber officinale var. rubrum (Rhizome extract) 80 mg
  * Foeniculi vulgare Fructus (Fennel) 25 mg
  * Menthae arvensis Folium (Mint) 5 mg
  * Piper retrofractum Fructus (Javanese long pepper) 12.5 mg
  * Honey 7500 mg
  Arms: Intervention Group (BEJO Red Ginger Extract)
Other: Placebo — Placebo composition: Substance without active ingredient
  Arms: Control Group (Placebo)

SUMMARY:
This study is a randomized, double-blind, placebo-controlled clinical trial to investigate the safety and efficacy of BEJO Red Ginger in hospitalized adult (18 - 50 years old) COVID-19 patients with mild clinical manifestations.

Subjects will be screened during hospitalization. One hundred and sixty-eight patients with confirmed SARS-CoV-2 infection and meeting all criteria, will be recruited to receive either BEJO Red Ginger or placebo in addition to standard of care (SOC) in a 1:1 ratio.

Patients with a diagnosis of COVID-19 and, due to mild symptoms, hospitalized, will be randomized to take a sachet of syrups containing 15 ml of BEJO Red Ginger, 3 times a day: 1 sachet after breakfast, 1 sachet after lunch, and 1 sachet after dinner, as add-on to the SOC, with 2 hours of incubation of SOC. The treatment will last for 14 days or until patients to be declared as cured. The treated patients will be compared with an equal group treated with placebo and SOC. Recovery time, symptoms, and objective (inflammatory) parameters (see detailed description) will be analyzed as outcomes. The goal of this study is to evaluate the role of BEJO Red Ginger in preventing progression of COVID-19 and accelerating healing process in patients.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 to 50 years, both sexes.
* Newly diagnosed adult patients with positive SARS-COV-2 by Real Time-PCR, using an appropriate sample such as nasopharyngeal, oropharyngeal, or nasal swab (within 3 days prior to study enrolment).
* Patients diagnosed with mild clinical manifestations, according to the Management of COVID-19 patients issued by The Indonesian Society of Respirology (Kepmenkes HK.0107/MENKES/5671/2021). Mild symptoms including fever, cough, shortness of breath, myalgia, sore throat, anosmia, diarrhea, nauseous and other symptoms.
* Hospitalized patients.
* Subject must have provided written informed consent which includes signing the institutional review board approved consent form prior to participating.

Exclusion Criteria:

* Asymptomatic COVID-19 patients
* Presence of any of the following abnormal laboratory values:

  * Elevation in serum glutamic oxaloacetic transaminase (SGOT) and/ or serum glutamic pyruvic transaminase (SGPT) of greater than 5 times the upper limit of normal (SGOT normal value 34 - 45 UI; SGPT normal value 31 - 35 UI)
  * Elevation in urea and creatinine blood levels of greater than the upper limit of normal (Urea normal value 10 - 44 mg/dL; creatinine normal value 0.4 - 1.4 mg/dL)
* Patients with severe pneumonia.
* Patients with serious co-morbidity, including: coronary heart diseases, congestive heart failure, arrhythmia, liver diseases, hypertension, diabetes mellitus (DM) type 1 and 2, glucocorticoid-induced DM, geriatric syndromes, autoimmune diseases, severe renal impairment, myocardial infarction, chronic obstructive pulmonary diseases (including asthma, tuberculosis) , and malignancies. The medical history was determined by from the statement of prospective subjects.
* Patients with ST-segment elevation myocardial infarction (STEMI) and non-ST-segment elevation myocardial infarction (NSTEMI), proved by an electrocardiogram (ECG) result.
* Be pregnant, confirmed with a negative pregnancy test.
* Lactating and breast feeding.
* Has consumed, or consuming herbal medicines or supplements other than SOC for COVID-10 in RSDC Wisma Atlet.
* Patient who has allergies to the test product.
* Active participation in other drug clinical trials.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 168 (Estimated)
Dates: Start 2022-02-22 (Actual); Primary Completion 2022-07-22 (Estimated); Study Completion 2022-08-22 (Estimated)

PRIMARY OUTCOMES:
Nucleic acid conversion time from randomization to the date of negative RT-PCR test result on the determined examinations. | from randomization to day 14 or until hospital discharge

SECONDARY OUTCOMES:
Clinical improvement; from initiation of study treatment (active or placebo) and daily anamnesis. | from randomization to day 14 or until hospital discharge
  Time to clinical improvement, defined as the time from randomization to improvement of subjects' clinical status.
Assessment of IL-6 level | from randomization to day 14 or until hospital discharge
  Changes from baseline in IL-6
Assessment of TNF-alfa level | from randomization to day 14 or until hospital discharge
  Changes from baseline in TNF-alfa

OTHER OUTCOMES:
Incidence of adverse events (AEs) and clinical worsening in patients hospitalized with COVID-19 should be referred to referral hospital. | from randomization to day 14 or until hospital discharge
  Number of AEs and clinical worsening that are unusual, unexpected or assessed as related to the investigational product.
Biochemical assessment of serum SGOT level | from randomization to day 14 or until hospital discharge
  Concentration of serum SGOT level in I/U. Biochemical assessment is measured 2 times: at the baseline and hospital discharge or the first of negative RT-PCR test result.
Biochemical assessment of serum SGPT level | from randomization to day 14 or until hospital discharge
  Concentration of serum SGPT level in I/U. Biochemical assessment is measured 2 times: at the baseline and hospital discharge or the first of negative RT-PCR test result.
Biochemical assessment of urea level | from randomization to day 14 or until hospital discharge
  Concentration of urea level in mg/dl. Biochemical assessment is measured 2 times: at the baseline and hospital discharge or the first of negative RT-PCR test result.
Biochemical assessment of creatinine level | from randomization to day 14 or until hospital discharge
  Concentration of creatinine level in mg/dl. Biochemical assessment is measured 2 times: at the baseline and hospital discharge or the first of negative RT-PCR test result.
Peripheral blood smear test | from randomization to day 14 or until hospital discharge
  Assessment of blood cell count for diagnosis of Covid-19 associated inflammation.

CONTACTS AND LOCATIONS:
Overall Officials: Erlang Samoedro, MD, Principal Investigator — Persahabatan General Hospital; Intan Satwika Putri, S.T, M.T, Study Director — National Research and Innovation Agency of Indonesia; Putro Setyobudyo Muhammad, MD, Study Chair — RSDC Wisma Atlet
Locations (1):
- RSDC Wisma Atlet Kemayoran, Jakarta, Indonesia